CLINICAL TRIAL: NCT04679233
Title: Feasibility and Preliminary Efficacy of Aerobic Exercise in Head and Neck Cancer Patients Undergoing Radiation Therapy
Brief Title: Feasibility and Safety of Aerobic Exercise for Head and Neck Cancer Patients
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI has withdrawn from the program, the study never started.
Sponsor: Vanderbilt University (Other)
Collaborators: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 201579
Record Dates: First submitted 2020-11-25; First posted 2020-12-22 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Head and Neck Neoplasm; Radiotherapy
Keywords: Head and Neck Neoplasm; Radiotherapy; Exercise
MeSH Terms: conditions — Head and Neck Neoplasms; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single group pre-test, post-test feasibility and safety study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Arm 1: Intervention Arm (Experimental): Arm 1 will receive the aerobic prescription exercise intervention. As this is a feasibility and safety study, there will not be a second arm.
  Interventions: Other: Prescription aerobic exercise

INTERVENTIONS:
Other: Prescription aerobic exercise — high intensity interval training, 5 weeks, 2 sessions/week - supervised by a clinician.

SUMMARY:
Treated head and neck cancer patients are subject to tissue swelling and scarring, known as lymphedema and fibrosis (LEF). LEF in the head and neck cancer patient occurs in up to 90% of treated patients and is associated with inflammation cells. Aerobic exercise is known to mediate these same inflammatory cells in an anti-inflammatory manner due to chronic adaptation of the cells. The investigators are therefore proposing a prescription exercise study for head and neck cancer patients. This study's primary aim is feasibility and safety of the aerobic exercise prescription. Feasibility of gathering study participant inflammation markers, visible LEF, and patient LEF symptoms will be a secondary aim of the study. Patient will be asked to journal their experience for a qualitative analysis. The prescription aerobic exercise is that of high intensity interval exercise, since this form of exercise can achieve similar or better results to moderate exercise with less time and patient burden. Each exercise session will take place on a cycle ergometer, will be 5 minutes warm up, 5 minutes cool down, and 20 minutes of exercise (1 minute intervals alternated by 1 minute rests x 10 each).

DETAILED DESCRIPTION:
Treated head and neck cancer patients are subject to tissue swelling and scarring, known as lymphedema and fibrosis (LEF). LEF in the head and neck cancer patient occurs in up to 90% of treated patients, is associated with inflammation cells. Aerobic exercise is known to mediate these same inflammatory cells in an anti-inflammatory manner due to chronic adaptation of the cells. The investigators are therefore proposing a prescription exercise study for head and neck cancer patients. This study's primary aim is feasibility and safety. Feasibility of gathering study participant inflammation markers, visible LEF, and patient LEF symptoms will be a secondary aim of the study. Patient will be asked to journal their experience for a qualitative analysis.

Based on the evidence, the aerobic exercise prescription for those who provide informed consent will consist of 10 intervals of intensity, and 10 intervals at rest. Each interval of intensity will be 1 minutes long and each rest period will be 1 minute long, and there will be a five-minute warm-up and five-minute cool down of easy pedaling for a total of 30 minutes. Participants will complete two sessions per week, and there will be at least one business day in between each session, for a total of 10 total exercise sessions. The total study duration will be less than 35 days.

The supervised prescribed HIIE intervention will be performed on a stationary cycle ergometer. A cycle ergometer is preferred for safety reasons since it requires less gross motor coordination than might be required with a treadmill. To assist in establishing safety (primary aim), the study participants heart rate will be continually monitored by a clinician during the exercise, guiding them to keep their heart rate within their specifically calculated 80-95% of their maximum HR during the periods of intensity.

The investigators will compare outcomes at baseline with outcomes at the end of the 5-week study period.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age
* Histologic proof of primary diagnosis of head and neck cancer
* Follow routinely with primary care doctor/general practitioner as evidenced by proof of appointment within the last 24 months)
* Ability to understand English in order to understand instructions and complete questionnaires
* Willing to participate in the supervised exercise intervention
* In the planning stages of/or actively receiving IMRT
* Must sign study-specific informed consent
* Medical clearance by attending physician

Exclusion Criteria:

* Evidence of distant metastasis prior to enrollment
* Simultaneous primaries or unknown primary
* Medical conditions that would prohibit the safe implementation of a an aerobic exercise practice per ACSM guidelines: cardiovascular disease, pulmonary disease, metabolic disease, or renal disease or signs/symptoms suggestive of cardiovascular disease at rest or during activity which include pain, discomfort in the chest, neck (other than caused by malignancy), jaw, arms, or other areas that may result from ischemia; shortness of breath at rest or with mild exertion; dizziness or syncope; orthopnea or paroxysmal nocturnal dyspnea; ankle edema; palpitations or tachycardia; intermittent claudication; known heart murmur; or unusual fatigue or shortness of breath with usual activities
* An answer of "no" on any of the Physical Activity Readiness Questionnaire (PAR-Q+) screening questions
* Pregnant or lactating women

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-02 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Qualitative Feasibility Log of Recruitment of Participants | 6 months
  To assess the feasibility of recruitment of a prescribed HIIE aerobic exercise modality for HNC patients. This will be measured by a Researchers Log which will include qualitative information regarding noted barriers to recruitment and reasons for patients not participating
Quantified and Qualitative Log of Feasibility of Implementation | 6 months
  To investigate the feasibility of a prescribed HIIE aerobic exercise modality for HNC patients. This will be measured by a Researchers Log which will include reasons that participants may have missed any of their assigned exercise sessions, as well as how many times they missed it.
Quantified and Qualitative Retention Log of Participants | 6 months
  To assess retention of a prescribed HIIE aerobic exercise modality for HNC patient. This will be measured by a Researchers Log which will include information such as number of participants enrolled, number of participants who dropped out, and reason for drop-out if available
Safety of the intervention as noted by parameters for serum bloodwork | 6 months
  To determine the safety of a prescribed HIIE aerobic exercise modality for HNC patients. This will be measured by a Researchers Log to ensure predetermined labs and electrolytes (platelets, magnesium, phosphorus, potassium) are within study parameter limits each week.
Safety of the intervention as noted by parameters for vitals signs prior to participation | 6 months
  To determine the safety of a prescribed HIIE aerobic exercise modality for HNC patients. This will be measured by a Researchers Log which will include ensuring vitals signs (heart rate in beats per minute, blood pressure in mmHg, oxygen in saturation, respiration rate in rate per minutes, and temperature in celsius) are within study parameter limits
Safety of the intervention as noted by a timely log of adverse events, | 6 months
  To determine the safety of a prescribed HIIE aerobic exercise modality for HNC patients. This will be measured by a Researchers Log which will include information such as measured by the CTCAE adverse events reported in accordance with and to the IRB

SECONDARY OUTCOMES:
Feasibility of Collecting Bloodwork - Biomarker MMP-9 | 6 months
  To assess the feasibility of collecting and using biomarkers as an outcome measure for research on the efficacy of a supervised prescribed HIIE modality for HNC patients. Collection of the following biomarkers is proposed: MMP-9. This will be measured as a blood draw, measured as ng/ml. Feasibility will be dichotomized and assessed as "yes" or "no" collected at both time points. Feasibility will be defined as 80% of blood draws collected at prescribed time.
Feasibility of Collecting Bloodwork at two time points - Biomarker IL-6 | 6 months
  To assess the feasibility of collecting and using biomarkers as an outcome measure for research on the efficacy of a supervised prescribed HIIE modality for HNC patients. Collection of the following biomarkers is proposed: IL-6. This will be measured as a blood draw, measured as pg/ml. Feasibility will be dichotomized and assessed as "yes" or "no" collected at both time points. Feasibility will be defined as 80% of blood draws collected at prescribed time.
Feasibility of Collecting Bloodwork at two time points - Biomarker IL-1β | 6 months
  To assess the feasibility of collecting and using biomarkers as an outcome measure for research on the efficacy of a supervised prescribed HIIE modality for HNC patients. Collection of the following biomarkers is proposed: IL-1β. This will be measured as a blood draw, measured as pg/ml. Feasibility will be dichotomized and assessed as "yes" or "no" collected at both time points. Feasibility will be defined as 80% of blood draws collected at prescribed time.
Feasibility of Collecting Bloodwork at two time points - Biomarker TNF-α | 6 months
  To assess the feasibility of collecting and using biomarkers as an outcome measure for research on the efficacy of a supervised prescribed HIIE modality for HNC patients. Collection of the following biomarkers is proposed: TNF-α. This will be measured as a blood draw, measured as pg/ml. Feasibility will be dichotomized and assessed as "yes" or "no" collected at both time points. Feasibility will be defined as 80% of blood draws collected at prescribed time.
Feasibility of Collecting Bloodwork at two time points - TGF-β1 | 6 months
  To assess the feasibility of collecting and using biomarkers as an outcome measure for research on the efficacy of a supervised prescribed HIIE modality for HNC patients. Collection of the following biomarkers is proposed: TGF-β1. This will be measured as a blood draw, measured as ng/mL. Feasibility will be dichotomized and assessed as "yes" or "no" collected at both time points. Feasibility will be defined as 80% of blood draws collected at prescribed time.
Feasibility of Collecting Patient Reported Outcome at two time points | 6 months
  To establish the feasibility of collecting the following outcome during the supervised prescribed HIIE regiment: LEF-related patient reported symptoms. The measurement tool to be used will be a validated a reliable patient reported outcome tool called the Lymphedema Symptom Inventory Distress Screening (LSIDS). Feasibility will be dichotomized and assessed as "yes" or "no" collected at both time points. Feasibility will be defined as 80% of LSIDS questionnaires completed in full.
Feasibility of Clinician Outcome at two time points | 6 months
  To establish the feasibility of collecting the following outcome during the supervised prescribed HIIE regiment: External Swelling LEF. The measurement tool to be used will be a standardized, validated, and reliable digital photography technique. Feasibility will be dichotomized and assessed as "yes" or "no" collected at both time points. Feasibility will be defined as 80% of digital photographs were able to be collected at prescribed time. Those with < 80% completed will be categorized as "no"
Qualitative data on Patient Experience | 6 months
  To gather preliminary feedback on the impact of a supervised prescribed HIIE regimen on patient perceived experience of the weekly exercise program as they undergo treatment via the measurement instrument of a personal and de-identified patient journal with self guided questions for patients to respond to open-endedly. This is to be analyzed qualitatively via qualitative content analysis

CONTACTS AND LOCATIONS:
Overall Officials: Bethany Rhoten, PhD, Study Chair — Vanderbilt University
Locations (1):
- Johns Hopkins, Baltimore, Maryland, United States

IPD SHARING:
Plan to Share IPD: No
individual participant data will not be shared. It will be de-identified prior to analysis.

REFERENCES:
- [Background] Nelson ME, Rejeski WJ, Blair SN, Duncan PW, Judge JO, King AC, Macera CA, Castaneda-Sceppa C. Physical activity and public health in older adults: recommendation from the American College of Sports Medicine and the American Heart Association. Med Sci Sports Exerc. 2007 Aug;39(8):1435-45. doi: 10.1249/mss.0b013e3180616aa2. PMID 17762378
- [Background] Schmitz KH, Courneya KS, Matthews C, Demark-Wahnefried W, Galvao DA, Pinto BM, Irwin ML, Wolin KY, Segal RJ, Lucia A, Schneider CM, von Gruenigen VE, Schwartz AL; American College of Sports Medicine. American College of Sports Medicine roundtable on exercise guidelines for cancer survivors. Med Sci Sports Exerc. 2010 Jul;42(7):1409-26. doi: 10.1249/MSS.0b013e3181e0c112. PMID 20559064
- [Background] Straub JM, New J, Hamilton CD, Lominska C, Shnayder Y, Thomas SM. Radiation-induced fibrosis: mechanisms and implications for therapy. J Cancer Res Clin Oncol. 2015 Nov;141(11):1985-94. doi: 10.1007/s00432-015-1974-6. Epub 2015 Apr 25. PMID 25910988
- [Background] Ridner SH, Dietrich MS, Sonis ST, Murphy B. Biomarkers Associated with Lymphedema and Fibrosis in Patients with Cancer of the Head and Neck. Lymphat Res Biol. 2018 Nov 28;16(6):516-24. doi: 10.1089/lrb.2017.0074. Online ahead of print. PMID 30484735
- [Background] Venkatesulu BP, Mahadevan LS, Aliru ML, Yang X, Bodd MH, Singh PK, Yusuf SW, Abe JI, Krishnan S. Radiation-Induced Endothelial Vascular Injury: A Review of Possible Mechanisms. JACC Basic Transl Sci. 2018 Aug 28;3(4):563-572. doi: 10.1016/j.jacbts.2018.01.014. eCollection 2018 Aug. PMID 30175280
- [Background] Ridner SH, Dietrich MS, Niermann K, Cmelak A, Mannion K, Murphy B. A Prospective Study of the Lymphedema and Fibrosis Continuum in Patients with Head and Neck Cancer. Lymphat Res Biol. 2016 Dec;14(4):198-205. doi: 10.1089/lrb.2016.0001. Epub 2016 Jun 15. PMID 27305456
- [Background] Elrefaey S, Massaro MA, Chiocca S, Chiesa F, Ansarin M. HPV in oropharyngeal cancer: the basics to know in clinical practice. Acta Otorhinolaryngol Ital. 2014 Oct;34(5):299-309. PMID 25709145
- [Background] Brayton KM, Hirsch AT, O Brien PJ, Cheville A, Karaca-Mandic P, Rockson SG. Lymphedema prevalence and treatment benefits in cancer: impact of a therapeutic intervention on health outcomes and costs. PLoS One. 2014 Dec 3;9(12):e114597. doi: 10.1371/journal.pone.0114597. eCollection 2014. PMID 25470383
- [Background] Brown M, McClean CM, Davison GW, Brown JCW, Murphy MH. The acute effects of walking exercise intensity on systemic cytokines and oxidative stress. Eur J Appl Physiol. 2018 Oct;118(10):2111-2120. doi: 10.1007/s00421-018-3930-z. Epub 2018 Jul 14. PMID 30008038
- [Background] Casuso RA, Aragon-Vela J, Huertas JR, Ruiz-Ariza A, Martinez-Lopez EJ. Comparison of the inflammatory and stress response between sprint interval swimming and running. Scand J Med Sci Sports. 2018 Apr;28(4):1371-1378. doi: 10.1111/sms.13046. Epub 2018 Jan 24. PMID 29281146
- [Background] Cullen T, Thomas AW, Webb R, Hughes MG. Interleukin-6 and associated cytokine responses to an acute bout of high-intensity interval exercise: the effect of exercise intensity and volume. Appl Physiol Nutr Metab. 2016 Aug;41(8):803-8. doi: 10.1139/apnm-2015-0640. Epub 2016 Mar 18. PMID 27377137
- [Background] Elmer DJ, Laird RH, Barberio MD, Pascoe DD. Inflammatory, lipid, and body composition responses to interval training or moderate aerobic training. Eur J Appl Physiol. 2016 Mar;116(3):601-9. doi: 10.1007/s00421-015-3308-4. Epub 2015 Dec 31. PMID 26721463
- [Background] Gmiat A, Micielska K, Kozlowska M, Flis DJ, Smaruj M, Kujach S, Jaworska J, Lipinska P, Ziemann E. The impact of a single bout of high intensity circuit training on myokines' concentrations and cognitive functions in women of different age. Physiol Behav. 2017 Oct 1;179:290-297. doi: 10.1016/j.physbeh.2017.07.004. Epub 2017 Jul 5. PMID 28687176
- [Background] Hoekstra SP, Bishop NC, Leicht CA. Can intervals enhance the inflammatory response and enjoyment in upper-body exercise? Eur J Appl Physiol. 2017 Jun;117(6):1155-1163. doi: 10.1007/s00421-017-3602-4. Epub 2017 Apr 4. PMID 28378071
- [Background] Hojman P, Brolin C, Norgaard-Christensen N, Dethlefsen C, Lauenborg B, Olsen CK, Abom MM, Krag T, Gehl J, Pedersen BK. IL-6 release from muscles during exercise is stimulated by lactate-dependent protease activity. Am J Physiol Endocrinol Metab. 2019 May 1;316(5):E940-E947. doi: 10.1152/ajpendo.00414.2018. Epub 2019 Feb 19. PMID 30779630
- [Background] van de Vyver M, Engelbrecht L, Smith C, Myburgh KH. Neutrophil and monocyte responses to downhill running: Intracellular contents of MPO, IL-6, IL-10, pstat3, and SOCS3. Scand J Med Sci Sports. 2016 Jun;26(6):638-47. doi: 10.1111/sms.12497. Epub 2015 Jun 9. PMID 26059973
- [Background] Ranadive SM, Kappus RM, Cook MD, Yan H, Lane AD, Woods JA, Wilund KR, Iwamoto G, Vanar V, Tandon R, Fernhall B. Effect of acute moderate exercise on induced inflammation and arterial function in older adults. Exp Physiol. 2014 Apr;99(4):729-39. doi: 10.1113/expphysiol.2013.077636. Epub 2014 Jan 24. PMID 24465022
- [Background] Zabihiyeganeh M, Vafaee Afshar S, Amini Kadijani A, Jafari D, Bagherifard A, Janbozorgi M, Akbari A, Mirzaei A. The effect of cognitive behavioral therapy on the circulating proinflammatory cytokines of fibromyalgia patients: A pilot controlled clinical trial. Gen Hosp Psychiatry. 2019 Mar-Apr;57:23-28. doi: 10.1016/j.genhosppsych.2019.01.003. Epub 2019 Jan 15. PMID 30669022
- [Background] Ostrowski K, Rohde T, Asp S, Schjerling P, Pedersen BK. Pro- and anti-inflammatory cytokine balance in strenuous exercise in humans. J Physiol. 1999 Feb 15;515 ( Pt 1)(Pt 1):287-91. doi: 10.1111/j.1469-7793.1999.287ad.x. PMID 9925898
- [Background] Zhang JM, An J. Cytokines, inflammation, and pain. Int Anesthesiol Clin. 2007 Spring;45(2):27-37. doi: 10.1097/AIA.0b013e318034194e. PMID 17426506
- [Background] Samuel SR, Maiya AG, Fernandes DJ, Guddattu V, Saxena PUP, Kurian JR, Lin PJ, Mustian KM. Effectiveness of exercise-based rehabilitation on functional capacity and quality of life in head and neck cancer patients receiving chemo-radiotherapy. Support Care Cancer. 2019 Oct;27(10):3913-3920. doi: 10.1007/s00520-019-04750-z. Epub 2019 Mar 27. PMID 30919154
- [Background] Adamsen L, Quist M, Andersen C, Moller T, Herrstedt J, Kronborg D, Baadsgaard MT, Vistisen K, Midtgaard J, Christiansen B, Stage M, Kronborg MT, Rorth M. Effect of a multimodal high intensity exercise intervention in cancer patients undergoing chemotherapy: randomised controlled trial. BMJ. 2009 Oct 13;339:b3410. doi: 10.1136/bmj.b3410. PMID 19826172
- [Background] Freitag N, Weber PD, Sanders TC, Schulz H, Bloch W, Schumann M. High-intensity interval training and hyperoxia during chemotherapy: A case report about the feasibility, safety and physical functioning in a colorectal cancer patient. Medicine (Baltimore). 2018 Jun;97(24):e11068. doi: 10.1097/MD.0000000000011068. PMID 29901612
- [Background] Adams SC, DeLorey DS, Davenport MH, Fairey AS, North S, Courneya KS. Effects of high-intensity interval training on fatigue and quality of life in testicular cancer survivors. Br J Cancer. 2018 May;118(10):1313-1321. doi: 10.1038/s41416-018-0044-7. Epub 2018 May 8. PMID 29736007
- [Background] Viana RB, de Lira CAB, Naves JPA, Coswig VS, Del Vecchio FB, Ramirez-Campillo R, Vieira CA, Gentil P. Can We Draw General Conclusions from Interval Training Studies? Sports Med. 2018 Sep;48(9):2001-2009. doi: 10.1007/s40279-018-0925-1. PMID 29675669
- [Background] Adlard KN, Jenkins DG, Salisbury CE, Bolam KA, Gomersall SR, Aitken JF, Chambers SK, Dunn JC, Courneya KS, Skinner TL. Peer support for the maintenance of physical activity and health in cancer survivors: the PEER trial - a study protocol of a randomised controlled trial. BMC Cancer. 2019 Jul 3;19(1):656. doi: 10.1186/s12885-019-5853-4. PMID 31269917
- [Background] Alizadeh S, Isanejad A, Sadighi S, Khalighfard S, Alizadeh AM. Effect of a high-intensity interval training on serum microRNA levels in women with breast cancer undergoing hormone therapy. A single-blind randomized trial. Ann Phys Rehabil Med. 2019 Sep;62(5):329-335. doi: 10.1016/j.rehab.2019.07.001. Epub 2019 Aug 7. PMID 31400480
- [Background] Baguley BJ, Skinner TL, Leveritt MD, Wright OR. Nutrition therapy with high intensity interval training to improve prostate cancer-related fatigue in men on androgen deprivation therapy: a study protocol. BMC Cancer. 2017 Jan 3;17(1):1. doi: 10.1186/s12885-016-3022-6. PMID 28049525
- [Background] Bhatia C, Kayser B. Preoperative high-intensity interval training is effective and safe in deconditioned patients with lung cancer: A randomized clinical trial. J Rehabil Med. 2019 Oct 3;51(9):712-718. doi: 10.2340/16501977-2592. PMID 31468059
- [Background] Boereboom CL, Blackwell JEM, Williams JP, Phillips BE, Lund JN. Short-term pre-operative high-intensity interval training does not improve fitness of colorectal cancer patients. Scand J Med Sci Sports. 2019 Sep;29(9):1383-1391. doi: 10.1111/sms.13460. Epub 2019 May 29. PMID 31116453
- [Background] Dasso NA. How is exercise different from physical activity? A concept analysis. Nurs Forum. 2019 Jan;54(1):45-52. doi: 10.1111/nuf.12296. Epub 2018 Oct 17. PMID 30332516
- [Background] Denlinger CS, Carlson RW, Are M, Baker KS, Davis E, Edge SB, Friedman DL, Goldman M, Jones L, King A, Kvale E, Langbaum TS, Ligibel JA, McCabe MS, McVary KT, Melisko M, Montoya JG, Mooney K, Morgan MA, O'Connor T, Paskett ED, Raza M, Syrjala KL, Urba SG, Wakabayashi MT, Zee P, McMillian N, Freedman-Cass D. Survivorship: introduction and definition. Clinical practice guidelines in oncology. J Natl Compr Canc Netw. 2014 Jan;12(1):34-45. doi: 10.6004/jnccn.2014.0005. PMID 24453291
- [Background] Devin JL, Sax AT, Hughes GI, Jenkins DG, Aitken JF, Chambers SK, Dunn JC, Bolam KA, Skinner TL. The influence of high-intensity compared with moderate-intensity exercise training on cardiorespiratory fitness and body composition in colorectal cancer survivors: a randomised controlled trial. J Cancer Surviv. 2016 Jun;10(3):467-79. doi: 10.1007/s11764-015-0490-7. Epub 2015 Oct 19. PMID 26482384
- [Background] Hwang CL, Yu CJ, Shih JY, Yang PC, Wu YT. Effects of exercise training on exercise capacity in patients with non-small cell lung cancer receiving targeted therapy. Support Care Cancer. 2012 Dec;20(12):3169-77. doi: 10.1007/s00520-012-1452-5. Epub 2012 Apr 14. PMID 22526147
- [Background] Kampshoff CS, Chinapaw MJ, Brug J, Twisk JW, Schep G, Nijziel MR, van Mechelen W, Buffart LM. Randomized controlled trial of the effects of high intensity and low-to-moderate intensity exercise on physical fitness and fatigue in cancer survivors: results of the Resistance and Endurance exercise After ChemoTherapy (REACT) study. BMC Med. 2015 Oct 29;13:275. doi: 10.1186/s12916-015-0513-2. PMID 26515383
- [Background] Lee K, Kang I, Mortimer JE, Sattler F, Mack WJ, Fitzsimons LA, Salem G, Dieli-Conwright CM. Effects of high-intensity interval training on vascular function in breast cancer survivors undergoing anthracycline chemotherapy: design of a pilot study. BMJ Open. 2018 Jun 30;8(6):e022622. doi: 10.1136/bmjopen-2018-022622. PMID 29961039
- [Background] Licker M, Karenovics W, Diaper J, Fresard I, Triponez F, Ellenberger C, Schorer R, Kayser B, Bridevaux PO. Short-Term Preoperative High-Intensity Interval Training in Patients Awaiting Lung Cancer Surgery: A Randomized Controlled Trial. J Thorac Oncol. 2017 Feb;12(2):323-333. doi: 10.1016/j.jtho.2016.09.125. Epub 2016 Oct 19. PMID 27771425
- [Background] Mijwel S, Bolam KA, Gerrevall J, Foukakis T, Wengstrom Y, Rundqvist H. Effects of Exercise on Chemotherapy Completion and Hospitalization Rates: The OptiTrain Breast Cancer Trial. Oncologist. 2020 Jan;25(1):23-32. doi: 10.1634/theoncologist.2019-0262. Epub 2019 Aug 7. PMID 31391297
- [Background] Midtgaard J, Christensen JF, Tolver A, Jones LW, Uth J, Rasmussen B, Tang L, Adamsen L, Rorth M. Efficacy of multimodal exercise-based rehabilitation on physical activity, cardiorespiratory fitness, and patient-reported outcomes in cancer survivors: a randomized, controlled trial. Ann Oncol. 2013 Sep;24(9):2267-73. doi: 10.1093/annonc/mdt185. Epub 2013 May 23. PMID 23704198
- [Background] Mugele H, Freitag N, Wilhelmi J, Yang Y, Cheng S, Bloch W, Schumann M. High-intensity interval training in the therapy and aftercare of cancer patients: a systematic review with meta-analysis. J Cancer Surviv. 2019 Apr;13(2):205-223. doi: 10.1007/s11764-019-00743-3. Epub 2019 Feb 26. PMID 30806875
- [Background] Oberste M, Schaffrath N, Schmidt K, Bloch W, Jager E, Steindorf K, Hartig P, Joisten N, Zimmer P. Protocol for the "Chemobrain in Motion - study" (CIM - study): a randomized placebo-controlled trial of the impact of a high-intensity interval endurance training on cancer related cognitive impairments in women with breast cancer receiving first-line chemotherapy. BMC Cancer. 2018 Nov 6;18(1):1071. doi: 10.1186/s12885-018-4992-3. PMID 30400840
- [Background] Papadopoulos E, Santa Mina D. Can we HIIT cancer if we attack inflammation? Cancer Causes Control. 2018 Jan;29(1):7-11. doi: 10.1007/s10552-017-0983-y. Epub 2017 Nov 21. PMID 29164363
- [Background] Schulz SVW, Laszlo R, Otto S, Prokopchuk D, Schumann U, Ebner F, Huober J, Steinacker JM. Feasibility and effects of a combined adjuvant high-intensity interval/strength training in breast cancer patients: a single-center pilot study. Disabil Rehabil. 2018 Jun;40(13):1501-1508. doi: 10.1080/09638288.2017.1300688. Epub 2017 Mar 21. PMID 28325109
- [Background] Schmitt J, Lindner N, Reuss-Borst M, Holmberg HC, Sperlich B. A 3-week multimodal intervention involving high-intensity interval training in female cancer survivors: a randomized controlled trial. Physiol Rep. 2016 Feb;4(3):e12693. doi: 10.14814/phy2.12693. PMID 26869680
- [Background] Schluter K, Schneider J, Sprave T, Wiskemann J, Rosenberger F. Feasibility of Two High-Intensity Interval Training Protocols in Cancer Survivors. Med Sci Sports Exerc. 2019 Dec;51(12):2443-2450. doi: 10.1249/MSS.0000000000002081. PMID 31730562
- [Background] Toohey K, Pumpa K, McKune A, Cooke J, DuBose KD, Yip D, Craft P, Semple S. Does low volume high-intensity interval training elicit superior benefits to continuous low to moderate-intensity training in cancer survivors? World J Clin Oncol. 2018 Feb 10;9(1):1-12. doi: 10.5306/wjco.v9.i1.1. PMID 29468132
- [Background] Thompson PD, Arena R, Riebe D, Pescatello LS; American College of Sports Medicine. ACSM's new preparticipation health screening recommendations from ACSM's guidelines for exercise testing and prescription, ninth edition. Curr Sports Med Rep. 2013 Jul-Aug;12(4):215-7. doi: 10.1249/JSR.0b013e31829a68cf. No abstract available. PMID 23851406
- [Background] Riebe D, Franklin BA, Thompson PD, Garber CE, Whitfield GP, Magal M, Pescatello LS. Updating ACSM's Recommendations for Exercise Preparticipation Health Screening. Med Sci Sports Exerc. 2015 Nov;47(11):2473-9. doi: 10.1249/MSS.0000000000000664. PMID 26473759
- [Background] Patterson JM, Hildreth A, Wilson JA. Measuring edema in irradiated head and neck cancer patients. Ann Otol Rhinol Laryngol. 2007 Aug;116(8):559-64. doi: 10.1177/000348940711600801. PMID 17847721
- [Background] Deng J, Dietrich MS, Murphy B. Self-care for head and neck cancer survivors with lymphedema and fibrosis: study protocol for a randomized controlled trial. Trials. 2019 Dec 27;20(1):775. doi: 10.1186/s13063-019-3819-0. PMID 31882012
- [Background] Dwivedi RC, St Rose S, Roe JW, Khan AS, Pepper C, Nutting CM, Clarke PM, Kerawala CJ, Rhys-Evans PH, Harrington KJ, Kazi R. Validation of the Sydney Swallow Questionnaire (SSQ) in a cohort of head and neck cancer patients. Oral Oncol. 2010 Apr;46(4):e10-4. doi: 10.1016/j.oraloncology.2010.02.004. Epub 2010 Mar 9. PMID 20219415
- [Background] List MA, D'Antonio LL, Cella DF, Siston A, Mumby P, Haraf D, Vokes E. The Performance Status Scale for Head and Neck Cancer Patients and the Functional Assessment of Cancer Therapy-Head and Neck Scale. A study of utility and validity. Cancer. 1996 Jun 1;77(11):2294-301. doi: 10.1002/(SICI)1097-0142(19960601)77:113.0.CO;2-S. PMID 8635098
- [Background] Ito S. High-intensity interval training for health benefits and care of cardiac diseases - The key to an efficient exercise protocol. World J Cardiol. 2019 Jul 26;11(7):171-188. doi: 10.4330/wjc.v11.i7.171. PMID 31565193
- [Background] Lanier JB, Mote MB, Clay EC. Evaluation and management of orthostatic hypotension. Am Fam Physician. 2011 Sep 1;84(5):527-36. PMID 21888303
- [Background] La Gerche A, Heidbuchel H. Can intensive exercise harm the heart? You can get too much of a good thing. Circulation. 2014 Sep 16;130(12):992-1002. doi: 10.1161/CIRCULATIONAHA.114.008141. No abstract available. PMID 25223770
- [Background] Lippi G, Sanchis-Gomar F. The health risks of acute exercise should also matter to internal medicine. Eur J Intern Med. 2011 Dec;22(6):e143. doi: 10.1016/j.ejim.2011.05.014. Epub 2011 Jul 7. No abstract available. PMID 22075302
- [Background] Guiraud T, Labrunee M, Gaucher-Cazalis K, Despas F, Meyer P, Bosquet L, Gales C, Vaccaro A, Bousquet M, Galinier M, Senard JM, Pathak A. High-intensity interval exercise improves vagal tone and decreases arrhythmias in chronic heart failure. Med Sci Sports Exerc. 2013 Oct;45(10):1861-7. doi: 10.1249/MSS.0b013e3182967559. PMID 23591293
- [Background] Lucini D, Pagani M. Exercise: Should it matter to internal medicine? Eur J Intern Med. 2011 Aug;22(4):363-70. doi: 10.1016/j.ejim.2011.02.022. Epub 2011 Mar 23. No abstract available. PMID 21767753
- [Background] Silver HJ, Dietrich MS, Murphy BA. Changes in body mass, energy balance, physical function, and inflammatory state in patients with locally advanced head and neck cancer treated with concurrent chemoradiation after low-dose induction chemotherapy. Head Neck. 2007 Oct;29(10):893-900. doi: 10.1002/hed.20607. PMID 17405169